CLINICAL TRIAL: NCT05066061
Title: Study of the Contribution of Virtual Reality Distraction in Peripheral Intravenous Catheter Insertion to Children From 6 to 11 Years in a Pediatric Day Hospital
Brief Title: Virtual Reality and Peripheral Intravenous Catheter Insertion to Children (R3VP)
Acronym: R3VP
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: recruiting difficulties
Sponsor: University Hospital, Clermont-Ferrand (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: AOI 2020 SAVEL; 2020-A03229-30 (Other: ANSM)
Record Dates: First submitted 2021-09-06; First posted 2021-10-04 (Actual); Last update posted 2025-11-20 (Actual); Status verified 2025-11

CONDITIONS: Virtual Reality; Catheterization, Peripheral Venous; Children, Only; Pain, Procedural
Keywords: virtual reality mask; children from 6 to 11; peripheral intravenous catheter insertion; pediatric's day hospital
MeSH Terms: conditions — Pain, Procedural | interventions — Anti-Anxiety Agents

STUDY DESIGN:
Intervention Model Description: Randomized, controlled, open-label, three-arm parallel, single-center therapeutic trial.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- standard (Active Comparator): Only use local anesthetic cream
  Interventions: Other: control arm
- anxiolytic gas (Experimental): Use local anesthetic cream and anesthetic and anxiolytic gas
  Interventions: Other: anxiolytic and analgesic gas
- virtual reality (Experimental): Use local anesthetic cream and virtual reality mask
  Interventions: Device: Virtual reality mask

INTERVENTIONS:
Other: control arm — usual process
  Arms: standard
Other: anxiolytic and analgesic gas — add relaxing gas
  Arms: anxiolytic gas
Device: Virtual reality mask — use Virtual reality mask Oculus Quest with age-appropriate software
  Arms: virtual reality

SUMMARY:
Main objective :

Evaluate the effect of using a virtual reality mask during the peripheral intravenous catheter insertion in a pediatric day hospital on the pain and anxiety in children from 6 to 11 years old.

Hypothesis :

Using virtual reality mask during the peripheral intravenous catheter insertion would reduce the 6 to 11 child's pain, the children and parents' anxiety, would improve satisfaction of children, parents and nurse about the care and would reduce time and cost of the procedure.

DETAILED DESCRIPTION:
Peripheral intravenous catheter insertion is a difficult, painful and anxiety-provoking procedure for hospitalized children, with the possible memorization of pain being even more present for children with chronic pathologies.

Memorization of painful events plays an essential role in anticipating the next experience and can lead to long-term consequences. The child, whose cognitive faculties are gradually developing and whose emotions are very invasive, is particularly concerned by this repercussion.

Different techniques can be used to prevent pain during care (apart from "human" techniques such as comfort, distraction by voice, information on gesture... which are part of good practice).

The national drug safety agency recommends the use of the local anesthetic cream and/or an equimolar mixture of oxygen and nitrous oxide causing surface anesthesia and relaxation and amnesia of the gesture.

Immersion in virtual reality allows to saturate the child's sensorially (3D vision, hearing and kinesthetic proprioception) thus reducing nociceptive perceptions and anxiety. His attention is focused by the virtual animation proposed during this experience. There are many devices (glasses, masks...) as well as various programs more or less specific to care situations, some of them allow to interact with games.

There is no randomized study comparing the efficacy on pain, satisfaction and anxiety of peripheral intravenous catheter insertion with the three possible analgesia techniques: local anesthetic cream / local anesthetic cream and anesthetic and anxiolytic gas / local anesthetic cream and virtual reality mask, nor on the medico-economic impact respecting standard 6 on homogeneous pediatric age groups in clinical trials.

This is a randomized, open-label, three-armed, parallel, single-center therapeutic trial comparing an analgesic strategy using two authorized medical devices (conventional strategy) with a virtual reality mask distraction technique for intravenous catheter insertion in children aged 6 to 11 years old hospitalized in the day hospital of Clermont Ferrand University Hospital.

The control arm is the local anesthetic cream arm, the experimental arms are the local anesthetic cream + anesthetic and anxiolytic gas arm on the one hand and the local anesthetic cream + virtual reality mask type Oculus quest® with interactive program on the other hand.

After informing and obtaining the consent of the child and his parents, will be measured the pain/anxiety/salivary cortisol/heart rate of the child; anxiety of the parents. The nurse evaluates the venous capital of the child then times the time of care and collects (among other things) the number of operators required. Immediately after the treatment, and then 15 to 30 minutes after the insertion will be measured the pain/anxiety/heart rate of the child; anxiety of the parents. The salivary cortisol at 20 minutes after catheter insertion will reflect the stress felt by the child during the procedure. Finally, the satisfaction of the child, parents, nurses will be collected 30 minutes after the care.

After statistical analysis of these three arms, it will be possible to determine the value of the anesthetic and anxiolytic gas and the virtual reality mask to reduce the child's pain and anxiety during the intravenous catheter insertion.

ELIGIBILITY:
Inclusion Criteria:

* Children from 6 to 11 years old requiring an intravenous catheter insertion in a pediatric day hospital at the Clermont Ferrand University Hospital.
* Subjects and their parents who were informed about the study and gave informed consent
* Subjects who have had local anesthetic cream for 1-5 hours at the puncture site
* On the first attempt to apply intravenous catheter on the day of inclusion
* Subjects and their parents able to use the self-report scales proposed in the study.

Exclusion Criteria:

Children from 6 to 11 :

* Having a modification of pain's integration (spina bifida for example)
* Having received an analgesic before the care
* Requiring contact isolation
* With a history of seizures or motion sickness
* Born very prematurely (< 28 SA)
* Presenting a contraindication to the use of the local anesthetic cream
* Presenting a contraindication to the use of the anesthetic and anxiolytic gas.
* Presenting a contraindication to the use of the virtual reality mask: heart disease, epilepsy, psychiatric illness (major anxiety, post traumatic stress syndrome)

Ages: 6 Years to 11 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 34 (Actual)
Dates: Start 2021-12-06 (Actual); Primary Completion 2025-11-03 (Actual); Study Completion 2025-11-03 (Actual)

PRIMARY OUTCOMES:
change from baseline child's pain at 30 minutes after the care | - Before the care - Immediately after the care - 15 to 30 minutes after the care
  self-evaluation of children's pain with the visual analog scale in vertical position quote from 0 to 10, 10 represents the worst pain we can feel

SECONDARY OUTCOMES:
change from baseline child's anxiety at 30 minutes after the care | -before the care -immediately after the care -15 to 30 minutes after the care
  self-evaluation of children's anxiety with numerical scale from 1 to 10 (10= worst score)
change from baseline heart rate at 30 minutes after the care | -before the care -immediately after the care -15 to 30 minutes after the care
  - Measure of heart rate (number of heartbeats in one minute)
change from baseline salivary cortisol at 30 minutes after the care | -before the care -15 to 30 minutes after the care
  - salivary cortisol : results in µg/l
change from baseline parents' anxiety at 30 minutes after the care | -before the care - immediately after the care - 15 to 30 minutes after the care
  self-evaluation of parents' anxiety with scale number from 0 to 10 (10= worst score)
evaluation of the care with satisfaction questionnaire | 30 minutes after the care
  satisfaction of the care for children, parents and nurses with satisfaction questionnaire for children : a score from 1 to 3 (3= best score, very satisfied) for parents and nurses : a score from 1 to 5 (5= best score, very satisfied)

CONTACTS AND LOCATIONS:
Overall Officials: EMMANUELLE LABRAISE, NURSE, Principal Investigator — ClermontFerrandUH
Locations (1):
- CHU de Clermont-Ferrand, Clermont-Ferrand, France

IPD SHARING:
Plan to Share IPD: No